CLINICAL TRIAL: NCT00240110
Title: Valproate Efficacy in Cocaine-Bipolar Comorbidity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ihsan Salloum, Professor of Psychiatry, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20070289; R01DA019992 (NIH); 05080018 (Other: NIDA); DPMCDA (Other: NIDA)
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Bipolar Disorder; Cocaine Dependence
Keywords: Bipolar; Cocaine; Comorbidity
MeSH Terms: conditions — Bipolar Disorder; Cocaine-Related Disorders | interventions — Valproic Acid; Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lithium carbonate add on Placebo (Placebo Comparator): Lithium carbonate started and stabilized then participants randomized to placebo
  Interventions: Drug: Placebo; Drug: Lithium Carbonate
- Lithium carbonate add on Valproate (Experimental): Lithium carbonate started and stabilized then participants randomized to Valproate
  Interventions: Drug: Valproate; Drug: Lithium Carbonate

INTERVENTIONS:
Drug: Valproate — Valproate with dose titration to achieve blood levels within the therapeutic range
  Other Names: Divalproex sodium
  Arms: Lithium carbonate add on Valproate
Drug: Placebo — Control arm
  Other Names: Placebo control
  Arms: Lithium carbonate add on Placebo
Drug: Lithium Carbonate — All participants were started and stabilized on lithium carbonate as a standard treatment for bipolar disorder
  Other Names: Standard treatment

SUMMARY:
This proposal will test the efficacy of a promising pharmacological approach for the treatment of comorbid cocaine dependence and bipolar disorder. We propose a randomized, double blind, placebo controlled 12-week trial to test the efficacy of Divalproex sodium (Valproate) plus treatment as usual compared to placebo plus treatment as usual in decreasing cocaine use and stabilizing mood symptoms among patients with comorbid cocaine dependence and bipolar disorder. Treatment as usual includes the use of lithium carbonate for mood stabilization plus supportive psychosocial treatment.

DETAILED DESCRIPTION:
Bipolar disorder has the highest rate of association with cocaine and other substance use disorders than any other major severe psychiatric syndrome. This comorbidity represents a major treatment challenge and is associated with severe disability, morbidity, and heightened risk for suicide.

The aims of this study are:

1. Examine the efficacy of valproate plus treatment as usual compared to placebo plus treatment as usual in decreasing cocaine use in patients with cocaine dependence and comorbid bipolar disorder.
2. Determine whether primary vs. secondary cocaine dependence, bipolar subtype (depressed vs. manic/mixed) and the presence of additional substance use disorders moderate the association between treatment and cocaine use outcome.
3. Assess the effects of medication compliance and mood symptoms as mediators of cocaine use outcome.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for cocaine dependence and a concurrent bipolar disorder

Exclusion Criteria:

* Schizophrenia, schizoaffective, and any non-bipolar psychotic disorder, unipolar major depression, primary anxiety disorder, mental retardation, and signs of impaired cognitive functioning.
* Current DSM-IV criteria for dependence on substances other than cocaine, alcohol, cannabis, nicotine, or caffeine
* Neurological conditions including epilepsy, history of brain injury, encephalitis, or any organic brain syndrome or documented focally abnormal EEG
* Medical conditions including severe cardiac, liver, kidney, or liver disease.
* Pregnancy
* Inability or unwillingness to use contraceptive methods
* Any medical condition or other reason that in the opinion of the investigator would prevent the subject from completing the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2006-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan M Salloum, MD, MPH, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Miller School of Medicine, Department of Psychiatry, Miami, Florida
  - University of Miami Miller School of Medicine, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salloum IM, Douaihy A, Cornelius JR, Kirisci L, Kelly TM, Hayes J. Divalproex utility in bipolar disorder with co-occurring cocaine dependence: a pilot study. Addict Behav. 2007 Feb;32(2):410-5. doi: 10.1016/j.addbeh.2006.05.007. Epub 2006 Jun 30. PMID 16814474

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: High screen failure for not meeting inclusion/exclusion criteria and for lost to follow-up during screening
Groups:
- Lithium Carbonate Add on Placebo: Lithium started and then participants randomized to placebo
- Lithium Carbonate Add on Valproate: Lithium carbonate started and participants randomized to valproate
Period: Overall Study
Arm/Group | Lithium Carbonate Add on Placebo | Lithium Carbonate Add on Valproate
Started | 13 | 13
Completed | 7 | 6
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Lithium Carbonate Add on Placebo: Lithium carbonate started with titration to achieve blood levels within the therapeutic range and then participants randomized to placebo
- Lithium Carbonate Add on Valproate: Lithium carbonate started with titration to achieve blood levels within the therapeutic range and then participants randomized to valproate
- Total: Total of all reporting groups
Arm/Group | Lithium Carbonate Add on Placebo | Lithium Carbonate Add on Valproate | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (7.4) | 44 (7.7) | 45.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percentage of Cocaine-abstinent Days
Description: Change from baseline in percentage of self-report cocaine-abstinent (non-use) days (difference in base percent values)
Time Frame: Week 12
Population: All subjects with available data after assignment to study medications
Measure: Mean (Standard Deviation); unit: percentage of days cocaine abstinent
Arm/Group | Lithium Carbonate Add on Placebo | Lithium Carbonate Add on Valproate
Number analyzed (Participants) | 11 | 12
percentage of days cocaine abstinent | 16.4 (29.7) | 14.5 (20.3)

2. Secondary Outcome: Change From Baseline in Percentage of Money Spent on Cocaine
Description: Change from baseline in percentage of the amount of money spent on cocaine
Time Frame: week 12
Population: All subjects with available data after assignment to study medications
Measure: Mean (Standard Deviation); unit: Percentage of Money Spent on Cocaine
Groups:
- Lithium Carbonate Add on Placebo: Open label lithium carbonate as standard treatment and double blinded placebo
- Lithium Carbonate Add on Valproate: Open label lithium carbonate as standard treatment and double blinded valproate
Arm/Group | Lithium Carbonate Add on Placebo | Lithium Carbonate Add on Valproate
Number analyzed (Participants) | 11 | 12
Percentage of Money Spent on Cocaine | -43.6 (58.4) | -34.9 (56.1)

ADVERSE EVENTS:
Groups:
- Lithium Carbonate Add on Placebo: Lithium carbonate as standard treatment add on double blind placebo
- Lithium Carbonate Add on Valproate: Lithium carbonate as standard treatment add on double blind valproate
Arm/Group | Lithium Carbonate Add on Placebo | Lithium Carbonate Add on Valproate
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/13
Other Adverse Events (participants affected / at risk) | 10/13 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate Add on Placebo (N=13) | Lithium Carbonate Add on Valproate (N=13)
Hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — worsening related to substance abuse (benzodiazepines and opioids) led to excessive sedation and admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lithium Carbonate Add on Placebo (N=13) | Lithium Carbonate Add on Valproate (N=13)
Headache (General disorders) | 4 | 3
Heart palpatation (Cardiac disorders) | 1 | 1
Nausea, diarrhea (Gastrointestinal disorders) | 6 | 6
Increased urination (Renal and urinary disorders) | 3 | 3
Back wrist pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Restless, sleepless (Psychiatric disorders) | 4 | 5
Fall (General disorders) | 0 | 2
sexual dysfunction (Reproductive system and breast disorders) | 1 | 1
increased menses (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No